CLINICAL TRIAL: NCT01471028
Title: A Randomized, Open-Label, Multicenter, Controlled Study to Assess Safety and Efficacy of ELAD in Subjects With Alcohol-Induced Liver Decompensation (AILD)
Brief Title: Assess Safety and Efficacy of ELAD (Extracorporeal Liver Assist System) in Subjects With Alcohol-Induced Liver Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-208
Record Dates: First submitted 2011-11-07; First posted 2011-11-11 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Acute Alcoholic Hepatitis
Keywords: Acute alcoholic hepatitis; alcoholic; hepatitis; liver
MeSH Terms: conditions — Hepatitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELAD Treatment (Experimental): This group will receive treatment with ELAD plus standard of care treatment.
  Interventions: Biological: ELAD treatment
- Standard of care (Control) (Other): This group will receive standard of care treatment as defined in the protocol.
  Interventions: Other: Standard of care (Control)

INTERVENTIONS:
Biological: ELAD treatment — ELAD treatment consists of treatment with an extracorporeal liver assist system.
  Other Names: ELAD
  Arms: ELAD Treatment
Other: Standard of care (Control) — Control receives standard medical treatment.
  Other Names: Standard of care as defined by the protocol
  Arms: Standard of care (Control)

SUMMARY:
The primary objective of the study is to evaluate safety and efficacy of ELAD® with respect to overall survival (OS) of subjects with a clinical diagnosis of alcohol-induced liver decompensation (AILD) up to at least Study Day 91, with follow-up Protocol VTI-208E providing additional survival data up to a maximum of 5 years that will be included, as available, through VTI-208 study termination (after the last surviving enrolled subject completes Study Day 91).

Secondary objectives are to determine the proportion of survivors at Study Days 28 and 91.

Exploratory objectives are to evaluate the ability of ELAD to stabilize liver function, measured using the Model for End Stage Liver Disease (MELD)-based time to progression (TTP) up to Study Day 91, and the proportion of progression-free survivors (PFS) up to Study Days 28 and 91. Progression is defined as death or the first observed increase of at least 5 points from End of Study Day 1 MELD score (for both the ELAD and Control groups) until at least 24 hours after the ELAD Treatment Period is ended (end of Day 7 for Controls) and up to both End of Study Days 28 and 91 following Randomization.

DETAILED DESCRIPTION:
Subjects randomized to the ELAD® group will receive treatment with ELAD® for a maximum of five (5) 24 hour periods as well as standard of care treatment.

Subjects randomized to the Control group will receive standard of care treatment throughout the study.

The ITT population includes all randomized subjects assigned to the group to which they were randomized, irrespective of actual treatment administered. Participant, Baseline Characteristics, and Outcome Measures used the ITT population. The safety population is defined as all subjects who are randomized based on actual treatment received. All serious adverse events and all non-serious adverse events analyses used the safety population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Total bilirubin ≥ 8 mg/dL;
* A clinical diagnosis of alcohol-induced liver decompensation (AILD), based upon evidence (by lab test, medical history, or family interview) of a clinical judgment of a temporal (6 weeks or less) and causal relationship between use of alcohol and this onset of symptoms;
* Subjects meeting inclusion criteria 1 through 3 will be classified as having either:

  a. Severe acute alcoholic hepatitis (AAH), with: i. Medical history of alcohol abuse; AND ii. Maddrey score of ≥ 32; AND iii. AAH documented by either:

  1. Confirmatory liver biopsy; OR 2. Two or more of the following:
  1. Hepatomegaly,
  2. AST > ALT,
  3. Ascites,
  4. Leukocytosis (WBC count above lab normal at site), OR

  b. Alcohol-induced decompensation of chronic liver disease that is not acute alcoholic hepatitis (as defined above), with: i. MELD score of 18-35; AND ii. Underlying chronic liver disease documented by:
  1. Liver biopsy, AND/OR
  2. Laboratory findings, AND/OR
  3. Medical history;
* Not eligible for liver transplant during this hospitalization;
* Subject or legally authorized representative must provide Informed Consent;
* Subject must be eligible for Standard of Care treatment as defined in the protocol.

Exclusion Criteria:

* Platelet count < 40,000/mm3;
* International Normalization Ratio (INR) > 3.5;
* MELD Score > 35;
* AST > 500 IU/L;
* Evidence of infection unresponsive to antibiotics;
* Evidence of reduction in total bilirubin of 20% or more in the previous 72 hours, if available. Bilirubin measurements must be taken at least 12 hours after any procedure known to artificially alter serum bilirubin (e.g., administration of packed red blood cells, plasma exchange);
* Evidence of hemodynamic instability as defined by the following:

  1. Systolic blood pressure < 90 mmHg with evidence of diminished perfusion unresponsive to fluid resuscitation and/or low-dose pressor support; OR
  2. Mean arterial pressure (MAP) < 60 mmHg with evidence of diminished perfusion unresponsive to fluid resuscitation and/or low-dose pressor support; OR
  3. Requirement for escalating doses of vasopressor support prior to Screening; OR
  4. Subject at maximum vasopressor dose at Screening;
* Evidence of active bleeding or of major hemorrhage defined as requiring ≥ 2 units packed red blood cells to maintain stable hemoglobin occurring within 48 hours of Screening;
* Clinical evidence of liver size reduction due to cirrhosis (liver size of the craniocaudal diameter (sagittal view) < 10 cm when measured on the mid clavicular line (or equivalent measurement) by ultrasound, or liver volume < 750 cc as determined by CT), unless Investigator interpretation of the clinical evidence indicates liver size of < 10 cm or volume < 750 cc is not considered reduced for the individual subject;
* Occlusive portal vein thrombosis impairing hepatopetal flow, or evidence of bile duct obstruction;
* Evidence by physical exam, history, or laboratory evaluation, of significant concomitant disease with expected life expectancy of less than 3 months, including, but not limited to:

  1. Severe acute or chronic cardiovascular, central nervous system, or pulmonary disease;
  2. Cancer that has metastasized or has not yet been treated;
* Subject has chronic end-stage renal disease requiring chronic hemodialysis for more than 8 weeks (not classified as hepatorenal syndrome);
* Subject has liver disease related to homozygous hemachromatosis, Wilson's Disease, has non-alcoholic fatty liver disease, or Budd-Chiari Syndrome;
* Pregnancy as determined by β-human chorionic gonadotropin (HCG) results, or lactation;
* Participation in another investigational drug, biologic, or device study within one month of enrollment, except for observational studies (the observational study setting should not affect safety and/or efficacy of the VTI-208 clinical trial);
* Previous liver transplant;
* Previous enrollment in the treatment phase of another ELAD trial (e.g. a subject is not disqualified from enrollment in VTI-208 if they were screened for VTI-210 but did not qualify for enrollment in the treatment phase of the study and therefore did not receive ELAD or Control treatment;
* Have a Do Not Resuscitate or a Do Not Intubate (DNR/DNI) directive (or such local equivalent) or any other Advanced Directive limiting Standard of Care in place (the DNR/DNI criterion is not applicable in the UK);
* Refusal to participate in the VTI-208E follow-up study;
* Inability to provide an address for home visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stange, MD, Study Director — Vital Therapies, Inc.; David J Reich, MD, Principal Investigator — PA - Drexel University College of Medicine; Ram Subramanian, MD, Principal Investigator — GA - Emory University Hospital; Lewis Teperman, MD, Principal Investigator — NY - New York University Langone Medical Center; Robert Brown, MD, Principal Investigator — NY - Columbia University Medical Center; Julie Thompson, MD, Principal Investigator — MN - University of Minnesota Medical Center - Twin Cities Campus; Paul Gaglio, MD, Principal Investigator — NY - Montefiore Medical Center; Linda Sher, MD, Principal Investigator — CA - Keck Hospital of University of Southern California; David Wolf, MD, Principal Investigator — NY - Westchester Medical Center; Parvez Mantry, MD, Principal Investigator — TX - Methodist Dallas Medical Center; Ali Al-Khafaji, MD, Principal Investigator — PA - University of Pittsburgh Medical Center; Marquis E Hart, MD, Principal Investigator — WA - Swedish Medical Center - Transplant Program; David Bernstein, MD, Principal Investigator — NY - North Shore University Hospital; Sumeet K Asrini, MD, Principal Investigator — TX - Baylor University Medical Center; Thomas Ardiles, MD, Principal Investigator — AZ - Maricopa Integrated Health System; Charles Landis, MD, Principal Investigator — WA - University of Washington - Harborview Medical Center; Rohit Satoskar, MD, Principal Investigator — DC - Georgetown University Hospital; Nikunj Shah, MD, Principal Investigator — IL - Rush University Medical Center; Brian Borg, MD, Principal Investigator — MS - University of Mississippi Medical Center; Alan Wigg, MD, Principal Investigator — South Australia - Flinders Medical Centre - Bedford Park; Gary Jeffrey, Principal Investigator — Western Australia - Sir Charles Gairdner Hospital - Nedlands; Lance L Stein, MD, Principal Investigator — GA - Piedmont Atlanta Hospital; Talal Adhami, MD, Principal Investigator — OH - Cleveland Clinic Foundation; Simona Rossi, MD, Principal Investigator — PA - Albert Einstein Medical Center; Anne McCune, MD, Principal Investigator — UK - Bristol - United Hospitals Bristol NHS Foundation Trust; Ahmed M Elsharkawy, MD, Principal Investigator — UK - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital; Andre Duarte-Rojo, MD, Principal Investigator — AR - University of Arkansas for Medical Sciences; Angel Alsina, MD, Principal Investigator — FL - Tampa General Hospital; Jag Sunderram, MD, Principal Investigator — NJ - Rutgers University Hospital; Geoffrey McCaughan, MD, Principal Investigator — Australia - Royal Prince Alfred Hospital - New South Wales; Raza Malik, MD, Principal Investigator — MA - Beth Israel Deaconess Medical Center; Juan Gallegos-Orozco, MD, Principal Investigator — UT - University of Utah Hospital; Tarek I Hassanein, MD, Principal Investigator — CA - Sharp Coronado Hospital; Shahid Habib, MD, Principal Investigator — AZ - University of Arizona Medical Center; Winfred W Williams, MD, Principal Investigator — MA - Massachusetts General Hospital; Pedram Enayati, MD, Principal Investigator — CA - Cedars-Sinai Medical Center; Michael Allison, MD, Principal Investigator — UK - England - Cambridge University Hospitals NHS Foundation Trust; Rajiv Jalan, MD, Principal Investigator — UK - England - Royal Free Hospital; Alexander Kuo, MD, Principal Investigator — CA - University of California San Diego Medical Center - Hillcrest; Alasdair Hay, MD, Principal Investigator — UK - Scotland - Royal Infirmary of Edinburgh; Agustin Albillos, MD, Principal Investigator — Spain - Madrid - Hospital Ramón y Cajal; Kalyan R Bhamidimarri, MD, Principal Investigator — FL - University of Miami Hospital; Xaralambos (Bobby) Zervos, DO, Principal Investigator — FL - Cleveland Clinic Florida; Waldo Concepcion, MD, Principal Investigator — CA - Stanford School of Medicine/Stanford University Medical Center; Julia A Wendon, MD, Principal Investigator — UK - England - King's College Hospital; Fred Poordad, MD, Principal Investigator — TX - The University of Texas Health Science Center - Texas Liver Institute
Locations (45):
- United States (35):
  - Maricopa Integrated Health System (MIHS), Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sharp Coronado Hospital, Coronado, California
  - Keck Hospital of University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford School of Medicine/Stanford University Medical Center, Palo Alto, California
  - University of California San Diego Medical Center - Hillcrest, San Diego, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota - Twin Cities Campus, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Rutgers University Hospital, New Brunswick, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas Health Science Center - Texas Liver Institute, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Swedish Medical Center - Transplant Program, Seattle, Washington
  - University of Washington - Harborview Medical Center, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Hospital Ramón y Cajal, Madrid, Spain
- United Kingdom (6):
  - King's College Hospital, London, England
  - Royal Free Hospital, Hamstead, London
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham, West Midlands
  - United Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh

REFERENCES:
- [Derived] Thompson J, Jones N, Al-Khafaji A, Malik S, Reich D, Munoz S, MacNicholas R, Hassanein T, Teperman L, Stein L, Duarte-Rojo A, Malik R, Adhami T, Asrani S, Shah N, Gaglio P, Duddempudi A, Borg B, Jalan R, Brown R, Patton H, Satoskar R, Rossi S, Parikh A, ElSharkawy A, Mantry P, Sher L, Wolf D, Hart M, Landis C, Wigg A, Habib S, McCaughan G, Colquhoun S, Henry A, Bedard P, Landeen L, Millis M, Ashley R, Frank W, Henry A, Stange J, Subramanian R; VTI-208 Study Group. Extracorporeal cellular therapy (ELAD) in severe alcoholic hepatitis: A multinational, prospective, controlled, randomized trial. Liver Transpl. 2018 Mar;24(3):380-393. doi: 10.1002/lt.24986. PMID 29171941
- See also: Vital Therapies, Inc. website — http://www.vitaltherapies.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ELAD Treatment: Participants randomized to the ELAD group received ELAD treatment plus protocol-directed Standard of Care (SOC) treatment for a period of up to 5 days followed by Standard of Care treatment through STudy Day 91.
- Standard of Care (Control): Participants randomized to the Control group received protocol-directed Standard of Care treatment in accord with AASLD and EASL guidelines for up to 91 days.
Period: VTI-208
Arm/Group | ELAD Treatment | Standard of Care (Control)
Started | 96 | 107
Completed | 56 | 63
Not Completed | 40 | 44
Not completed — Adverse Event | 39 | 41
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Period: VTI-208E
Arm/Group | ELAD Treatment | Standard of Care (Control)
Started | 56 | 63
Database Lock, 31 July 2015 | 56 | 63
Completed | 48 | 51
Not Completed | 8 | 12
Not completed — Death | 7 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- ELAD Treatment: Participants randomized to the ELAD group received ELAD treatment plus protocol-directed Standard of Care treatment for a period of up to 5 days followed by Standard of Care treatment through Study Day 91.
- Total: Total of all reporting groups
Arm/Group | ELAD Treatment | Standard of Care (Control) | Total
Number analyzed (Participants) | 96 | 107 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 104 | 198
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (9.06) | 44.8 (10.66) | 45.6 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 55 | 65 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 84 | 91 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 93 | 176
  United Kingdom | 6 | 6 | 12
  Australia | 7 | 8 | 15
Baseline MELD Score [Mean (Standard Deviation); unit: MELD Score] — The Model for End-stage Liver Disease (MELD) score is calculated by the following formula: MELD SCORE= 0.95 x LOGc (creatinine g/dL) + 0.378 x Logc (bilirubin mg/dL) + 1.120 x Logc (INR) + 0.643. The 3 tests, bilirubin (liver function), INR (blood clotting), and creatinine (kidney function), can all be affected by advanced liver disease. Scores range from 6 in a healthy person to 40, at which point a person is very sick and likely in a hospital ICU. MELD ≥28 typically indicates a poor outcome. Higher baseline MELD scores predict worse outcomes. In this study, the Min/Max MELD score was 20/35.
  MELD Score | 27.6 (3.94) | 27.1 (3.79) | 27.3 (3.86)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary endpoint of the study was a comparison of overall survival (OS) between the ELAD-treated and Control groups, with protocol VTI-208E providing additional survival data up to a maximum of 5 years, that was included as available at the time of database lock (31 July 2015).
Time Frame: Up to at least Study Day 91, with protocol VTI-208E providing additional survival data (at 6, 9, 12, 24 months) at the time of database lock (31 July 2015)
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD Treatment | Standard of Care (Control)
Number analyzed (Participants) | 96 | 107
Participants | 57 | 66
Statistical Analysis 1: Comparison: ELAD Treatment vs Standard of Care (Control); The primary endpoint was assessed using a Kaplan-Meier survival analysis of the Intent-to-treat (ITT) population utilizing a log-rank test; Test type: Superiority; p = 0.904, Log Rank; Hazard Ratio (HR) = 1.027, 95% CI 2-sided [0.689 to 1.53]

2. Secondary Outcome: Number of Survivors at Study Day 91.
Description: Assess the proportion of survivors at Study Day 91.
Time Frame: Up to Study Day 91.
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD Treatment | Standard of Care (Control)
Number analyzed (Participants) | 96 | 107
Participants | 57 | 66
Statistical Analysis 1: Comparison: ELAD Treatment vs Standard of Care (Control); Test type: Superiority; p = 0.737, Chi-squared

3. Other Pre Specified Outcome: Number of Progression-free Survivors at Study Day 91
Description: An exploratory objective is to evaluate the ability of ELAD® to stabilize liver function, measured using the MELD-based time to progression (TTP), with progression defined as death or the first observed increase of at least 5 points from End of Study Day 1 MELD score (for both the ELAD and Control groups) until at least 24 hours after the ELAD Treatment Period is ended (end of Day 7 for Controls) and up to both End of Study Days 28 and 91 following Randomization.
Time Frame: Study Day 1 up to Study Day 91
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD Treatment | Standard of Care (Control)
Number analyzed (Participants) | 96 | 107
Participants | 45 | 59
Statistical Analysis 1: Comparison: ELAD Treatment vs Standard of Care (Control); Test type: Superiority; p = 0.168, Log Rank; Hazard Ratio (HR) = 1.315, 95% CI 2-sided [0.886 to 1.952]

4. Post Hoc Outcome: Overall Survival for Subjects With Age<50, MELD<30, Bili>=16, INR<=2.5 and Creatinine<1.3
Description: Creatinine <1.3 INR <=2.5 Bilirubin >=16 Age <50 MELD <30
Time Frame: as for outcome 1
Population: Kaplan-Meier
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD Treatment | Standard of Care (Control)
Number analyzed (Participants) | 96 | 107
Participants | 29 | 31
Statistical Analysis 1: Comparison: ELAD Treatment vs Standard of Care (Control); Test type: Superiority; p = 0.007, Log Rank; Hazard Ratio (HR) = 0.283, 95% CI 2-sided [0.109 to 0.732]

ADVERSE EVENTS:
Time Frame: Randomization through Study Day 91.
Description: According to the SAP, Safety Population was used for the analysis of all adverse events and was defined according to the actual treatment received. Two subjects were not treated with ELAD because they did not meet the safety eligibility criteria and were included in the Control group. One subject who randomized to Control but received ELAD treatment and this subject was included in the ELAD group. Therefore, 95 subjects were exposed to ELAD treatment and 108 subjects were exposed to Control.
Arm/Group | ELAD Treatment | Standard of Care (Control)
All-Cause Mortality (participants affected / at risk) | 38/95 | 42/108
Serious Adverse Events (participants affected / at risk) | 73/95 | 75/108
Other Adverse Events (participants affected / at risk) | 95/95 | 107/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD Treatment (N=95) | Standard of Care (Control) (N=108)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytophenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis bacterial (Gastrointestinal disorders) | 2 (2) | 3 (3)
Alcohol withdrawal syndrome (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 7 (7) | 10 (10)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Ascites (Hepatobiliary disorders) | 6 (6) | 13 (16)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 8 (11) | 6 (7)
Hepatic failure (Hepatobiliary disorders) | 13 (14) | 10 (10)
Hepatitis alcoholic (Hepatobiliary disorders) | 2 (2) | 4 (4)
Hepatorenal syndrome (Hepatobiliary disorders) | 3 (4) | 9 (9)
Hyperammonaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (4)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Hepatotoxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (3) | 3 (6)
Generalised oedema (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delerium (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Emphysematous cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 12 (14)
Renal impairment (Renal and urinary disorders) | 2 (3) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Vascular disorders) | 7 (8) | 6 (6)
Haematochezia (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Myocardial infarction (Vascular disorders) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Vascular disorders) | 0 (0) | 1 (2)
Portal vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Vascular disorders) | 1 (1) | 3 (3)
Septic shock (Vascular disorders) | 2 (2) | 4 (4)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (Vascular disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD Treatment (N=95) | Standard of Care (Control) (N=108)
Anaemia (Blood and lymphatic system disorders) | 42 (47) | 17 (19)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anisocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 29 (34) | 13 (15)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypochromasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 13 (16) | 13 (13)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 33 (36) | 12 (12)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (6) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 4 (7)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 2 (2) | 1 (1)
Chest discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 7 (8) | 4 (4)
Dizziness (Vascular disorders) | 2 (3) | 12 (15)
Hyperdynamic left ventricle (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 0 (0)
Oedema peripheral (Metabolism and nutrition disorders) | 32 (38) | 33 (41)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Right atrial dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 7 (7) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 17 (19) | 10 (10)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (21) | 10 (12)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Dry Eye (Eye disorders) | 4 (4) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Keratopathy (Eye disorders) | 0 (0) | 1 (1)
Limbal swelling (Eye disorders) | 1 (1) | 0 (0)
Scleral discolouration (Eye disorders) | 0 (0) | 2 (2)
Scleral disorder (Eye disorders) | 1 (1) | 0 (0)
Scleral oedema (Eye disorders) | 2 (3) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 16 (17) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 27 (37) | 22 (29)
Abdominal tenderness (Gastrointestinal disorders) | 2 (3) | 3 (3)
Anastomotic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bacterascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 19 (20) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 19 (20) | 17 (19)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Faecal incontinence (Nervous system disorders) | 3 (3) | 3 (3)
Faeces discoloured (Gastrointestinal disorders) | 4 (4) | 4 (4)
Faeces pale (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (5) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 3 (3) | 2 (2)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Vascular disorders) | 6 (6) | 4 (5)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth haemorrhage (Vascular disorders) | 1 (1) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (18) | 23 (27)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oral discharge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 5 (5) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritoneal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis bacterial (Gastrointestinal disorders) | 6 (6) | 4 (4)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 4 (4)
Rectal haemorrhage (Vascular disorders) | 8 (9) | 4 (4)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 14 (17) | 17 (21)
Administration site pain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Asthenia (General disorders) | 6 (7) | 12 (14)
Catheter site haemorrhage (Injury, poisoning and procedural complications) | 9 (10) | 4 (4)
Cyst (General disorders) | 0 (0) | 2 (2)
Device component issue (General disorders) | 1 (1) | 0 (0)
Device damage (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Effusion (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 7 (7) | 6 (7)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Flank pain (General disorders) | 1 (1) | 1 (1)
Gait disturbance (Nervous system disorders) | 1 (1) | 3 (3)
Hyperthermia (General disorders) | 2 (2) | 0 (0)
Hypothermia (General disorders) | 3 (3) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Infusion site haemorrhage (General disorders) | 2 (2) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2)
Medical device complication (General disorders) | 2 (3) | 1 (1)
Mucosal dryness (General disorders) | 1 (1) | 2 (2)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 7 (8) | 9 (10)
Procedural pain (General disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 25 (28) | 10 (10)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Ascites (Hepatobiliary disorders) | 34 (37) | 30 (40)
Asterixis (Hepatobiliary disorders) | 9 (9) | 16 (16)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Caput medusae (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Coma hepatic (Nervous system disorders) | 2 (5) | 1 (1)
Foetor hepaticus (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 36 (45) | 29 (30)
Hepatic failure (Hepatobiliary disorders) | 2 (3) | 3 (3)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatorenal syndrome (Hepatobiliary disorders) | 11 (12) | 11 (13)
Hyperammonaemia (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hypoalbuminaemia (Hepatobiliary disorders) | 4 (4) | 7 (7)
Jaundice (Hepatobiliary disorders) | 2 (2) | 4 (4)
Ocular icterus (Hepatobiliary disorders) | 1 (1) | 3 (3)
Portal hypertension (Hepatobiliary disorders) | 2 (2) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 16 (18) | 7 (8)
Candidiasis (Infections and infestations) | 9 (10) | 3 (3)
Candiduria (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 4 (4) | 6 (6)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 2 (2) | 2 (2)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 3 (3) | 2 (2)
Fungal skin infection (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 8 (8) | 6 (6)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 10 (10)
Propionibacterium infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 7 (8)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 14 (19) | 16 (19)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Catheter site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Catheter site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Catheter site related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 5 (7)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Feeding tube complicaiton (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injection site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Vessel puncture site haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acinetobacter test positive (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alpha 1 foetoprotein increased (Investigations) | 2 (2) | 2 (3)
Ammonia abnormal (Investigations) | 0 (0) | 1 (1)
Ammonia increased (Investigations) | 3 (3) | 1 (1)
Antibiotic resistant Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 0 (0)
Aspiration bronchial (Investigations) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 5 (5) | 1 (1)
Blood aldosterone decreased (Investigations) | 0 (0) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood cortisol decreased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 4 (4)
Blood fibrinogen decreased (Investigations) | 4 (4) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 6 (6) | 1 (1)
Blood lactic acid abnormal (Investigations) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 4 (4) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 1 (1)
Blood phosphorous abnormal (Investigations) | 0 (0) | 1 (1)
Blood phosphorous decreased (Investigations) | 1 (1) | 1 (1)
Blood potassium abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Body surface area increased (Investigations) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 6 (6) | 4 (4)
Cardiac murmur (Investigations) | 10 (10) | 8 (10)
Clostridium test positive (Investigations) | 2 (2) | 1 (1)
Computerised tomogram head (Investigations) | 1 (1) | 0 (0)
Culture urine positive (Investigations) | 1 (1) | 2 (2)
Drug screen positive (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QRS complex abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 2 (2)
Enterococcus test positive (Investigations) | 1 (1) | 0 (0)
Full blood count abnormal (Investigations) | 1 (1) | 0 (0)
Fungal test positive (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (5) | 2 (2)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2) | 2 (2)
Procalcitonin increased (Investigations) | 2 (2) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (2) | 2 (2)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1)
Sputum culture positive (Investigations) | 3 (3) | 0 (0)
Total lung capacity decreased (Investigations) | 2 (2) | 0 (0)
Urine colour abnormal (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 4 (4) | 0 (0)
Volume blood decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 5 (6)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Generalised oedema (Metabolism and nutrition disorders) | 9 (9) | 4 (4)
Goitre (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (8) | 4 (6)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 6 (7) | 3 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 18 (24) | 3 (5)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (23) | 29 (34)
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 (25) | 14 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 15 (17)
Hypophasphataemia (Metabolism and nutrition disorders) | 23 (23) | 14 (14)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Lactic acidosis (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Localised oedema (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Metabolic acidosis (Metabolism and nutrition disorders) | 16 (16) | 13 (14)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Oedema (Metabolism and nutrition disorders) | 9 (9) | 12 (15)
Osteoporosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Zinc deficiency (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 13 (16)
Chills (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle atrophy (Nervous system disorders) | 8 (8) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stifness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (5)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colonic polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 16 (17) | 8 (8)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (2) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 14 (14) | 3 (3)
Convulsion (Nervous system disorders) | 2 (2) | 2 (3)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Facial spasm (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 11 (14) | 7 (7)
Hereditary cerebral degeneration (Nervous system disorders) | 2 (2) | 0 (0)
Hyperreflexia (Nervous system disorders) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 1 (1)
Hyporeflexia (Nervous system disorders) | 1 (1) | 0 (0)
Hyporesponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 14 (14) | 15 (15)
Lethargy (Nervous system disorders) | 4 (4) | 5 (5)
Mobility decreased (Nervous system disorders) | 2 (2) | 0 (0)
Muscular weakness (Nervous system disorders) | 1 (1) | 3 (3)
Myoclonic epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (2)
Nystagmus (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2) | 3 (3)
Pupils unequal (Nervous system disorders) | 1 (1) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 5 (5)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 14 (14) | 10 (11)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Amnesia (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 21 (22) | 9 (10)
Apraxia (Psychiatric disorders) | 1 (1) | 0 (0)
Catatonia (Psychiatric disorders) | 0 (0) | 1 (1)
Circadian rhythm sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 2 (2) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 7 (7)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (2)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Failure to thrive (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 3 (3) | 2 (2)
Hallucination, auditory (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Hypophagia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Korsakoff's syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Memory impairment (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (4) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Selective mutism (Psychiatric disorders) | 0 (0) | 1 (1)
Speech disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stupor (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Anuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 3 (3)
Costovertebral angle tenderness (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 4 (4) | 0 (0)
Micturation urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 6 (6) | 0 (0)
Polyuria (Renal and urinary disorders) | 4 (4) | 2 (2)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 22 (23) | 21 (25)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic calcification (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal irritation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (2) | 4 (4)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 6 (6)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (25) | 21 (26)
Epistaxis (Vascular disorders) | 10 (11) | 6 (6)
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngitis bacterial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 14 (14)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (5)
Rales (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anogenital warts (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Ecchymosis (Vascular disorders) | 9 (9) | 6 (9)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Eschar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Face oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial wasting (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Herpes simplex (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Onychomycosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Palmar erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Perianal erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 19 (20) | 19 (20)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 11 (12)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scratch (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Biliary drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Extubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Intravenous catheter management (Surgical and medical procedures) | 4 (4) | 0 (0)
Removal of foreign body from external ear (Surgical and medical procedures) | 0 (0) | 1 (1)
Suture insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal compartment syndrome (Vascular disorders) | 2 (2) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Vascular disorders) | 1 (1) | 0 (0)
Cardiovascular deconditioning (Vascular disorders) | 1 (1) | 0 (0)
Contusion (Vascular disorders) | 8 (8) | 6 (6)
Coronary artery disease (Vascular disorders) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Dizziness postural (Vascular disorders) | 2 (2) | 1 (1)
Gastric haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Gastric varices (Vascular disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Vascular disorders) | 4 (4) | 4 (4)
Gingival bleeding (Vascular disorders) | 1 (1) | 1 (1)
Haematochezia (Vascular disorders) | 3 (3) | 4 (4)
Haematoma (Vascular disorders) | 6 (6) | 3 (3)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemoptysis (Vascular disorders) | 3 (3) | 2 (2)
Haemorrhage (Vascular disorders) | 4 (5) | 0 (0)
Haemorrhage intracranial (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhoids (Vascular disorders) | 5 (5) | 8 (8)
Haemothorax (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 29 (37) | 18 (20)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0)
Melaena (Vascular disorders) | 5 (6) | 3 (4)
Mucosal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0)
Penile haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Petechiae (Vascular disorders) | 4 (5) | 2 (2)
Pharyngeal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Portal hypertensive gastropathy (Vascular disorders) | 3 (3) | 9 (9)
Portal vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Presyncope (Vascular disorders) | 0 (0) | 1 (1)
Procedural haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Vascular disorders) | 5 (5) | 0 (0)
Pulmonary hypertension (Vascular disorders) | 4 (4) | 0 (0)
Purpura (Vascular disorders) | 0 (0) | 3 (3)
Retroperitoneal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Scrotal haematoma (Vascular disorders) | 0 (0) | 1 (1)
Septic shock (Vascular disorders) | 5 (5) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Spider naevus (Vascular disorders) | 5 (5) | 5 (5)
Splenic infarction (Vascular disorders) | 0 (0) | 1 (1)
Splenic varices (Vascular disorders) | 0 (0) | 1 (1)
Splenic vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Syncope (Vascular disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (Vascular disorders) | 2 (2) | 3 (3)
Telangiectasia (Vascular disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Urogenital haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Vascular disorders) | 3 (3) | 1 (1)
Varices oesophageal (Vascular disorders) | 3 (3) | 6 (6)
Vascular anomaly (Vascular disorders) | 2 (2) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes